CLINICAL TRIAL: NCT01590628
Title: Allogeneic Stem Cell Transplantation of NiCord®, Umbilical Cord Blood-Derived Ex Vivo Expanded Stem and Progenitor Cells, in Patients With Hemoglobinopathies
Brief Title: Allogeneic SCT of NiCord®, UCB-Derived Ex Vivo Expanded Stem and Progenitor Cells, in Patients With Hemoglobinopathies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gamida Cell ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC P#02.01.020
Record Dates: First submitted 2012-04-15; First posted 2012-05-03 (Estimated); Results first posted 2022-04-27 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-04

CONDITIONS: Sickle Cell Disease & Thalassemia
Keywords: Sickle Cell Disease & Thalassemia; Genetic disorder
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NiCord (Experimental): NiCord: NiCord® is a cell-based product composed of umbilical cord-derived ex vivo expanded stem and progenitor cells.
  Interventions: Drug: NiCord

INTERVENTIONS:
Drug: NiCord — NiCord® is a cell-based product composed of umbilical cord-derived ex vivo expanded stem and progenitor cells

SUMMARY:
Allogeneic Stem Cell Transplantation of NiCord®, Umbilical Cord Blood-Derived Ex Vivo Expanded Stem and Progenitor Cells, in Patients with Hemoglobinopathies

DETAILED DESCRIPTION:
Umbilical cord blood (UCB) is an alternative stem cell source for hematopoietic stem cell transplantations (HSCT) and can be used for the treatment of various life-threatening diseases, such as hematological malignancies or genetic blood disorders, in such cases where a matched related stem cell donor is not available. However, the major drawback of using this valuable stem cells source is the limited cell dose in a single cord blood unit (CBU), which was shown to be associated with inadequate hematopoietic reconstitution and high risk of transplant-related mortality. To improve outcomes and extend applicability of UCB transplantation, one potential solution is ex vivo expansion of UCB-derived stem and progenitor cells. NiCord® is a stem/progenitor cell based product composed of ex vivo expanded allogeneic UCB cells. NiCord® is based on a novel technology for the ex vivo cell expansion of cord blood derived hematopoietic progenitor cells. By increasing the number of the short and long-term reconstitution progenitor cells transplanted, NiCord® has the potential to enable the broader application of UCB transplantation, and improve the clinical outcomes of UCB transplantation.

In Part 1 of this study, NiCord® will be administered to the patient in conjunction with a second, unmanipulated CBU. In Part 2 of this study, NiCord® will be administered to the patient without a second, unmanipulated CBU. The study duration per patient is approximately 270 days from signing of informed consent to last visit on day 180 post-transplant.

The overall study objectives of part 1 of this study are to evaluate the safety and efficacy of co-transplantation of NiCord® and an unmanipulated CBU in patients with Hemoglobinopathies (Sickle Cell Disease (SCD), or thalassemia major) following myeloablative therapy. The overall study objectives of part 2 of this study are to evaluate the safety and efficacy of transplantation of NiCord® in patients with Hemoglobinopathies (Sickle Cell Disease (SCD), or thalassemia major) following myeloablative therapy.

The study hypothesis for part 1 of this study is that the co-transplantation of NiCord® and an unmanipulated unrelated cord blood graft in patients with hemoglobinopathies (SCD, or thalassemia major) following myeloablative preparative therapy will be safe and will enable cord blood engraftment. The study hypothesis for part 2 of this study is that transplantation of NiCord® in patients with hemoglobinopathies (SCD, or thalassemia major) following myeloablative preparative therapy will be safe and will enable cord blood engraftment.

Up to fifteen (15) evaluable patients recruited for part 1 of the study and up to five (5) patients for part 2 of the study should be 2-45 years of age, at least 10 kg in weight, have symptomatic SCD or thalassemia major and should be considered as candidates for allogeneic myeloablative HSCT for the treatment of SCD.

ELIGIBILITY:
Inclusion Criteria:

* Must be 2 - 45 years of age and at least 10 kg
* Must have clinically severe SCD (SS, SC or SBeta0 Thal) or thalassemia major and be eligible for myeloablative SCT
* Must have two partially HLA-matched CBUs for part 1; and one partially HLA-matched CBU for part 2
* Back-up autologous stem cells harvested from bone marrow
* Adequate Karnofsky Performance score or Lansky Play-Performance scale
* Sufficient physiological reserves
* Signed written informed consent

Exclusion Criteria:

* HLA-matched related donor able to donate
* Severe alloimmunization with inability to guarantee a supply of adequate PRBC donors
* Prior allogeneic hematopoietic SCT within the last 12 months or reduced-intensity transplant within the past 6 months
* Human immunodeficiency virus (HIV) infection
* Active or uncontrolled infection
* Pregnancy or lactation

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University Medical Center, NC, USA; Joel Brochstein, MD, Principal Investigator — Steven & Alexandra Cohen Children's Medical Center, New York
Locations (3):
- United States (3):
  - Steven & Alexandra Cohen Children's Medical Center, New York, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The University Of Texas M. D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Parikh S, Brochstein JA, Galamidi E, Schwarzbach A, Kurtzberg J. Allogeneic stem cell transplantation with omidubicel in sickle cell disease. Blood Adv. 2021 Feb 9;5(3):843-852. doi: 10.1182/bloodadvances.2020003248. PMID 33560399
- See also: Duke University Medical Center — http://www.dukehealth.org/
- See also: Gamida Cell Ltd. — http://www.gamida-cell.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled and treated 16 patients in total. 13 patients were treated with omidubicel and an unmanipulated CBU and these served as the primary analysis population for all study endpoints. Three additional patients who were exposed to omidubicel as a single graft source, were included in the safety summaries in order to encompass the entire population exposed to omidubicel.
Groups:
- NiCord + Unmanipulated CBU: NiCord: NiCord® is a cell-based product composed of umbilical cord-derived ex vivo expanded stem and progenitor cells. NiCord was transplanted in Part 1 subjects, together with an unmanipulated CBU.
- NiCord: NiCord: NiCord® is a cell-based product composed of umbilical cord-derived ex vivo expanded stem and progenitor cells. NiCord was transplanted in Part 2 subjects as a standalone graft.
Period: Overall Study
Arm/Group | NiCord + Unmanipulated CBU | NiCord
Started | 13 | 3
Completed | 11 | 3
Not Completed | 2 | 0
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- NiCord + Unmanipulated CBU: NiCord: NiCord® is a cell-based product composed of umbilical cord-derived ex vivo expanded stem and progenitor cells.
  The NiCord was transplanted together with an unmanipulated CBU graft.
- NiCord: NiCord: NiCord® is a cell-based product composed of umbilical cord-derived ex vivo expanded stem and progenitor cells.
  The NiCord was transplanted as a standalone product.
- Total: Total of all reporting groups
Arm/Group | NiCord + Unmanipulated CBU | NiCord | Total
Number analyzed (Participants) | 13 | 3 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 3 | 16
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 1 | 10
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 3 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 3 | 16
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 3 | 16
Sickle Cell or Thalassemia Disease Type [Count of Participants; unit: Participants]
  Hb SS | 13 | 2 | 15
  Hb SC | 0 | 0 | 0
  Hb SBeta0 Thal | 0 | 1 | 1
  Hb SD | 0 | 0 | 0
  Hb SOarab | 0 | 0 | 0
  Other SCD Type | 0 | 0 | 0
  Beta Thal Major | 0 | 0 | 0
  Alpha Thal Major | 0 | 0 | 0
CMV Screen (IgG or Total) (Segment S) positive [Count of Participants; unit: Participants] | 7 | 2 | 9
Performance Status [Count of Participants; unit: Participants] — The Karnofsky Performance Scale Index allows patients to be classified as to their functional impairment on a scale of 0 to 100%. This can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. The lower the Karnofsky score, the worse the survival for most serious illnesses.
  Participants
    100 | 6 | 2 | 8
    90 | 3 | 0 | 3
    80 | 4 | 0 | 4
    70 | 0 | 1 | 1
Disease characteristics [Number; unit: participants]
  Three or More Recurrent Painful Events in the Past 2 Years | 6 | 2 | 8
  Acute Chest Syndrome (Two or More Episodes in the Past 2 Years) | 2 | 0 | 2
  SCD-related & clinically significant neurologic event | 4 | 1 | 5
  Abnormal MRI/MRA | 5 | 1 | 6
  chronic PRBC transfusion therapy | 0 | 0 | 0
  Patient has undergone TCD velocity tests | 1 | 0 | 1
Hydroxyurea use prior to enrollment [Count of Participants; unit: Participants] | 10 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Will be Measured by Acute NiCord® Infusional Toxicity.
Description: Assessment of acute toxicity associated with the infusion of NiCord within 24 hours post-infusion.
Time Frame: 24 hours post-infusion
Measure: Number; unit: participants
Groups:
- NiCord + Unmanipulated CBU: Participants who received NiCord together with an unmanipulated CBU.
- NiCord: Participants who received NiCord as a standalone graft.
Arm/Group | NiCord + Unmanipulated CBU | NiCord
Number analyzed (Participants) | 13 | 3
participants
  Grade 4-5 acute toxicity event | 0 | 0
  Grade 3 acute toxicity event | 3 | 0

2. Primary Outcome: Assessment of Cumulative Incidence of Donor-derived Neutrophil Engraftment.
Description: Neutrophil engraftment is defined as achieving an absolute neutrophil count (ANC) of ≥500/ μL for 3 consecutive measurements on different days by Day 42 inclusive (the day of engraftment was defined as the first of these 3 days).
Time Frame: By Day 42
Measure: Count of Participants; unit: Participants
Groups:
- NiCord as a Standalone Graft: NiCord was transplanted as a stand-alone graft in subjects that participated in Part 2.
Arm/Group | NiCord + Unmanipulated CBU | NiCord as a Standalone Graft
Number analyzed (Participants) | 13 | 3
Participants | 13 | 3

3. Secondary Outcome: Proportion of Transplant-related Mortality.
Description: Transplant-related mortality is defined as death not preceded by autologous recovery.
Time Frame: at 100 days
Measure: Number; unit: percentage of participants
Arm/Group | NiCord + Unmanipulated CBU | NiCord
Number analyzed (Participants) | 13 | 3
percentage of participants | 0 | 0

4. Secondary Outcome: Event-free Survival
Description: Patients with event-free survival at 100 days post-transplant that did not have one of the following events: death, autologous recovery, primary or secondary graft failure.
Time Frame: 100 days post-transplant
Population: In the first group, 13 patients received NiCord together with a second unmanipulated CBU. In the 2nd group, 3 patients received NiCord as a standalone graft. No statistical analysis was performed for this outcome as this number of patients is too small for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NiCord + Unmanipulated CBU | NiCord as a Standalone Graft
Number analyzed (Participants) | 13 | 3
percentage of participants | 92.3 [56.6 to 98.9] | 66.6 [NA to NA] — No statistical analysis was performed for this outcome as this number of patients is too small for analysis.

5. Secondary Outcome: Overall Survival
Description: Overall survival at 180 days
Time Frame: 180 days
Population: In the first group, 13 patients received NiCord together with a second unmanipulated CBU. In the 2nd group, 3 patients received NiCord as a standalone graft.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NiCord + Unmanipulated CBU | NiCord as a Standalone Graft
Number analyzed (Participants) | 13 | 3
percentage of participants | 92.3 [56.6 to 98.9] | 100 [NA to NA] — Due to the insufficient number of patients who received a standalone NiCord transplant (3 in total), no statistical anlysis was performed.

ADVERSE EVENTS:
Time Frame: adverse event data were collected throughout the post-transplant period (180 days) and 6 months post study completion (1 year post transplantation).
Groups:
- NiCord + Unmanipulated CBU: NiCord: NiCord® is a cell-based product composed of umbilical cord-derived ex vivo expanded stem and progenitor cells.
  The primary safety objective was to assess the acute toxicity associated with the infusion of omidubicel within 24 hours post-infusion.
  Part 1: The primary efficacy objective of Part 1 was to assess the cumulative incidence of donor-derived neutrophil engraftment by Day 42 following co-transplantation of omidubicel and unmanipulated cord blood grafts.
- NiCord: NiCord: NiCord® is a cell-based product composed of umbilical cord-derived ex vivo expanded stem and progenitor cells.
  The primary safety objective was to assess the acute toxicity associated with the infusion of omidubicel within 24 hours post-infusion.
  Part 2: The primary efficacy objective of Part 2 was to assess the cumulative incidence of donor-derived neutrophil engraftment by Day 42 following transplantation of single unit omidubicel.
Arm/Group | NiCord + Unmanipulated CBU | NiCord
All-Cause Mortality (participants affected / at risk) | 2/13 | 0/3
Serious Adverse Events (participants affected / at risk) | 13/13 | 3/3
Other Adverse Events (participants affected / at risk) | 0/13 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NiCord + Unmanipulated CBU (N=13) | NiCord (N=3)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Acute graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Graft versus host disease (Immune system disorders) | 3 (3) | 0 (0)
Transplant rejection (Immune system disorders) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 3 (3) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT01590628/Prot_SAP_000.pdf